CLINICAL TRIAL: NCT01682772
Title: A Phase II Trial of Olaparib in Patients With Advanced Castration Resistant Prostate Cancer (TOPARP)
Brief Title: TOPARP: A Phase II Trial of Olaparib in Patients With Advanced Castration Resistant Prostate Cancer
Acronym: TOPARP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2011/10030; 2011-000601-49 (EudraCT Number); CRUK/C12540/A12354 (Other Grant/Funding Number: Cancer Research UK); ISRCTN15124653 (Registry Identifier: Randomised Controlled Trials); ISS22810018 (Other Grant/Funding Number: Astra Zeneca)
Record Dates: First submitted 2012-07-27; First posted 2012-09-11 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: Olaparib; Adenocarcinoma; Prostate
MeSH Terms: conditions — Adenocarcinoma | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olaparib 400mg (Experimental): Oral Olaparib at a dose of 400mg twice daily, continuously on a 28 day cycle
  Interventions: Drug: Olaparib
- Olaparib 300mg (Experimental): Oral Olaparib at a dose of 300mg twice daily, continuously on a 28 day cycle
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Until objective disease progression, unacceptable toxicity or patient withdrawal for whatever reason
  Other Names: AZD2281

SUMMARY:
This is an open-label, single arm, two part adaptive design phase II trial of Olaparib in patients with advanced castration resistant prostate cancer.

The trial aims to evaluate the the anti-tumour activity of Olaparib in metastatic castration resistant prostate cancer, identify molecular signatures of tumour cells in responding and non-responding patients, and to identify predictive biomarkers of Olaparib response.

DETAILED DESCRIPTION:
Patients with advanced castration resistant prostate cancer will receive single agent Olaparib at a dose of 400mg twice daily, continuously on a 28 day cycle. Olaparib will be administered until objective disease progression or unacceptable toxicity or patient withdrawal for whatever reason

ELIGIBILITY:
Inclusion Criteria:

1. Subject capable of understanding & complying with protocol requirements & signed the informed consent form
2. Minimum age 18 years
3. Histologically confirmed adenocarcinoma of the prostate with tumour tissue available for molecular analyses
4. At least one but no more than two previous taxane-based chemotherapy regimens. If docetaxel chemotherapy is used more than once, this will be considered as one regime. Patients may have had prior exposure to cabazitaxel treatment
5. At least 28 days since the completion of prior therapy, including major surgery, chemotherapy & other investigational agents. Clinically relevant sequelae should have resolved to grade 1 or less prior to recommencing treatment. For hormonal treatment & radiotherapy refer to the protocol guidelines
6. Documented prostate cancer progression as described in the protocol.
7. Surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 2.0 nM). If the patient is being treated with LHRH agonists this must have been initiated at least 4 weeks prior to Cycle 1 Day 1 & must be continued throughout the study.
8. Eastern Cooperative Oncology Group Performance Status of 0, 1, 2
9. Life expectancy > 12 weeks
10. Able to swallow a whole tablet
11. Patient & the patient's partner of childbearing potential, must agree to use medically accepted methods of contraception during the course of the study & for 3 months after the last dose of study drug
12. Agreeable to have all the biomarker studies including the paired fresh tumour biopsies.
13. CTC count of 5 cells/7.5mls blood or more at screening. Note: For Part B, CTC count >5 cells/7.5mls blood is not mandatory if patient has measurable disease by modified RECIST and a lesion >2cm and PSA greater than or equal to 2ng/ml at screening.
14. Adequate bone marrow, hepatic & renal function as defined in the protocol
15. For Part B only, patients must have genomic defects associated with olaparib sensitivity identified by NGS by the central lab.

Exclusion Criteria:

1. Surgery, or local prostatic intervention (excluding a prostatic biopsy) less than 28 days of Cycle 1 Day 1
2. Less than 28 days from any active anticancer therapy or investigational agents. For hormonal treatment & radiotherapy refer to the guidelines outlined in the inclusion criteria
3. Prior treatment with a PARP inhibitor, platinum, cyclophosphamide or mitoxantrone chemotherapy
4. Uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV heart disease), unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension or psychiatric illness/social situations that would limit compliance with study requirements
5. Any acute toxicities due to prior chemotherapy & / or radiotherapy that have not resolved to a NCI-CTCAE v4.02 grade 0 or 1 with the exception of chemotherapy induced alopecia & grade 2 peripheral neuropathy
6. Malignancy within the previous 2-years with a > 30% probability of recurrence within 12 months with the exception of non-melanoma skin cancer, in-situ or superficial bladder cancer
7. Patients with myelodysplastic syndrome/acute myeloid leukaemia
8. Patients with known symptomatic brain metastasis are not suitable for enrollment. Patients with asymptomatic, stable, treated brain metastases are eligible for study entry
9. Patients with symptomatic or impending cord compression unless appropriately treated beforehand & clinically stable & asymptomatic
10. Patients who have experienced a seizure or seizures within 6 months of study treatment or who are currently being treated with cytochrome P450 enzyme inducing anti-epileptic drugs for seizures
11. Patients receiving any of the following classes of inhibitors of CYP3A4 (see protocol for guidelines & wash out periods)
12. Patients with gastrointestinal disorders likely to interfere with absorption of the study medication
13. Initiating bisphosphonate therapy or adjusting bisphosphonate dose/regimen within 30 days prior to Cycle 1 Day 1. Patients on a stable bisphosphonate regimen are eligible & may continue
14. Presence of a condition or situation, which, may put the patient at significant risk, confound the study results, or interfere significantly with participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Response rate to Olaparib | Response will be evaluated 6 months post trial entry
  Response will be defined on the basis of the following outcomes, if any of these occur patients will be considered to have responded:
  * Objective response by modified RECIST
  * PSA decline of ≥50% according to the Prostate Cancer Working Group 2
  * Conversion of circulating tumour cell count from ≥5 cells/7.5ml blood at baseline to <5 cells/7.5ml blood confirmed by at least two readings 4 weeks apart

SECONDARY OUTCOMES:
Radiographic progression free survival | Radiographic progression free survival will be evaluated 6 months post trial entry
  rPFS will be defined by either RECIST progression and/or progression on bone scan. It will be measured from the date of trial entry to the first occurence of radiographic progression or death from any cause
Progression free survival | Progression free survival will be evaluated 6 months post trial entry
  PFS will be measured from date of trial entry until radiographic progression, unequivocal clinical progression or death
Time to PSA Progression | Time to PSA progression will be evaluated 6 months post trial entry
  For patients who have achieved ≥50% decrease from the cycle 1 day 1 (baseline), the PSA progression date is defined as the date that a ≥25% increase and an absolute increase of ≥2ng.mL above the nadir is documented. This must be confirmed by a second consecutive value. For patients without a PSA decrease of this magnitude or no decrease at all, PSA progression date is defined as the date that a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the baseline is documented. This must also be confirmed by a second consecutive value.
CTC count conversion rate | CTC count conversion rate will be evaluated 6 months post trial entry
  Proportion of patients with conversion of CTC count from ≥5/7.5ml blood at baseline to <5/7.5ml blood nadir
Duration of PSA response | Duration of PSA response will be evaluated 6 months post trial entry
  Duration of PSA response is calculated from the time the PSA value first declines by at least 50% of the cycle 1 day 1 (baseline) value (must be confirmed by a second value) until the time there is an increase of 25% of PSA nadir, provided the absolute increase is at least 2 ng/mL. The increase must be confirmed by a second consecutive measurement.
Number of participants with grade 3 or 4 adverse events as a measure of safety and tolerability. | Will be evaluated 1) when the first 5 and 10 participants have completed the 1st cycle of treatment and, 2) at 6 months post trial entry.
  The proportion of patients with grade 3/4 adverse events will be described along with other descriptive measures of safety and tolerability and evaluated by the IDMC
Time to radiographic progression | Will be evaluated 6 months post trial entry
  Time to radiographic progression (progression defined by either RECIST progression and /or progression on bone scan) will be measured from the date of trial entry to the first occurrence of radiographic progression. Death from prostate cancer or any other cause without prior radiographic evidence of progression will not count as an event.
Overall survival | Will be evaluated 6 months post trial entry
  OS will be measured from the date of trial entry to the date of death (whatever the cause). Survival time of living patients will be censored on the last date a patient is known to be alive or lost to follow-up
PSA objective response | Will be evaluated 6 months post trial entry
  PSA response and PSA progression are defined according to the consensus guidelines of the Prostate Cancer Clinical Trials Working Group 2.

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (2):
- United Kingdom (2):
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - University College Hospital London, London

REFERENCES:
- [Derived] Carmichael J, Figueiredo I, Gurel B, Beije N, Yuan W, Rekowski J, Seed G, Carreira S, Bertan C, Fenor de La Maza MLD, Chandran K, Neeb A, Welti J, Gallagher L, Bogdan D, Crespo M, Riisnaes R, Ferreira A, Miranda S, Lu J, Shen MM, Hall E, Porta N, Westaby D, Guo C, Grochot R, Lord CJ, Mateo J, Sharp A, de Bono J. RNASEH2B loss and PARP inhibition in advanced prostate cancer. J Clin Invest. 2024 Jun 4;134(21):e178278. doi: 10.1172/JCI178278. PMID 38833311
- [Derived] Mateo J, Porta N, Bianchini D, McGovern U, Elliott T, Jones R, Syndikus I, Ralph C, Jain S, Varughese M, Parikh O, Crabb S, Robinson A, McLaren D, Birtle A, Tanguay J, Miranda S, Figueiredo I, Seed G, Bertan C, Flohr P, Ebbs B, Rescigno P, Fowler G, Ferreira A, Riisnaes R, Pereira R, Curcean A, Chandler R, Clarke M, Gurel B, Crespo M, Nava Rodrigues D, Sandhu S, Espinasse A, Chatfield P, Tunariu N, Yuan W, Hall E, Carreira S, de Bono JS. Olaparib in patients with metastatic castration-resistant prostate cancer with DNA repair gene aberrations (TOPARP-B): a multicentre, open-label, randomised, phase 2 trial. Lancet Oncol. 2020 Jan;21(1):162-174. doi: 10.1016/S1470-2045(19)30684-9. Epub 2019 Dec 2. PMID 31806540
- [Derived] Mateo J, Carreira S, Sandhu S, Miranda S, Mossop H, Perez-Lopez R, Nava Rodrigues D, Robinson D, Omlin A, Tunariu N, Boysen G, Porta N, Flohr P, Gillman A, Figueiredo I, Paulding C, Seed G, Jain S, Ralph C, Protheroe A, Hussain S, Jones R, Elliott T, McGovern U, Bianchini D, Goodall J, Zafeiriou Z, Williamson CT, Ferraldeschi R, Riisnaes R, Ebbs B, Fowler G, Roda D, Yuan W, Wu YM, Cao X, Brough R, Pemberton H, A'Hern R, Swain A, Kunju LP, Eeles R, Attard G, Lord CJ, Ashworth A, Rubin MA, Knudsen KE, Feng FY, Chinnaiyan AM, Hall E, de Bono JS. DNA-Repair Defects and Olaparib in Metastatic Prostate Cancer. N Engl J Med. 2015 Oct 29;373(18):1697-708. doi: 10.1056/NEJMoa1506859. PMID 26510020